CLINICAL TRIAL: NCT05472259
Title: A Non-comparative Randomized Phase 2 Study, Evaluating the Efficacy of 5-FU + NALIRI and 5-FU + NALIRINOX for Metastatic Pancreatic Ductal Adenocarcinoma (PDAC), Progressive After Gemcitabine-Abraxane or Gemcitabine Monotherapy
Brief Title: A Study Evaluating the Efficacy of 5-FU + NALIRI and 5-FU + NALIRINOX for PDAC (NALPAC)
Acronym: NALPAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Belgian Group of Digestive Oncology (Other)
Collaborators: University Hospital St Luc, Brussels (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NALPAC
Record Dates: First submitted 2021-12-09; First posted 2022-07-25 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A NALIRI (Active Comparator): Cycle length: 14 days
  Day 1:
  * Leucovorin: 400 mg/m² IV - Dilute in 250 mL DSW and administer over two hours
  * Liposomal irinotecan (FBE): 70 mg/m² IV* - Dilute in 500 mL DSW and administer over 90 min
  * 5 FU: 2400 mg/m² IV - Dilute in 500 to 1000 mL 0,9% NS of DSW and administer as a continuous IV infusion over 46 hours. To accommodate an ambulatory pump for outpatient treatment can be administered undiluted (50 mg/mL) or the total dose diluted in 100 to 150 mL NS.
    * Patients who are known to be homozygous for UGT1A1*28 should start treatment with 50 mg/m2 ONIVYDE. If they do not encounter drug related toxicities during the first cycle of therapy (started at a reduced dose of 50 mg/m2), they may have the dose of ONIVYDE increased to a dose of 70 mg/m2 in subsequent cycles based on individual patient tolerance.
  Interventions: Drug: Nanoliposomal irinotecan; Drug: 5 FU; Drug: Leucovorin
- Arm B NALIRINOX (Experimental): Cycle length: 14 days
  Day 1:
  * Oxaliplatin 60 mg IV - Dilute in 500 mL D5W and administer over two hours (prior to leucovorin). Shorter oxaliplatin administration schedules (eg. 1mg/m2 per minute) appear to be safe.
  * Leucovorin: 400 mg/m² IV - Dilute in 250 mL DSW and administer over two hours (after oxaliplatin)
  * Nanoliposomal irinotecan (FBE): 50 mg/m² IV - Dilute in 500 mL D5W and administer over 90 min
  * 5 FU: 2400 mg/m² IV - Dilute in 500 to 1000 mL 0,9% NS of DSW and administer as a continuous IV infusion over 46 hours. To accommodate an ambulatory pump for outpatient treatment can be administered undiluted (50 mg/mL) or the total dose diluted in 100 to 150 mL NS.
  Interventions: Drug: Nanoliposomal irinotecan; Drug: 5 FU; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Nanoliposomal irinotecan — In the control arm (Naliri) a dose of 70mg/m² is administered in combination with 5FU and leucovorin In the investigational arm (Nalirinox) a dose of 50mg/m² is administered in combination with 5FU, leucovorin and oxaliplatin
  Other Names: Onyvide
Drug: 5 FU — In the control arm (Naliri) a dose of 2400 mg/m² is administered in combination with nanoliposomal irinotecan and leucovorin In the investigational arm (Nalirinox) a dose of 2400 mg/m² is administered in combination with nanoliposomal irinotecan, leucovorin and oxaliplatin
  Other Names: Fluorouracil
Drug: Leucovorin — In the control arm (Naliri) a dose of 400 mg/m² is administered in combination with nanoliposomal irinotecan and 5FU In the investigational arm (Nalirinox) a dose of 400 mg/m² is administered in combination with nanoliposomal irinotecan, 5FU and oxaliplatin
  Other Names: Folinate; Elvorine
Drug: Oxaliplatin — Only administered in the investigational arm (Nalirinox): a dose of 60 mg/m² is administered in combination with nanoliposomal irinotecan, 5FU and Leucovorin
  Arms: Arm B NALIRINOX

SUMMARY:
A non-comparative randomized phase 2 study, evaluating the efficacy of 5-FU + NALIRI and 5-FU + NALIRINOX for metastatic pancreatic ductal adenocarcinoma (PDAC), progressive after Gemcitabine-Abraxane or Gemcitabine monotherapy

DETAILED DESCRIPTION:
Based on the results of previous studies, the sponsor aims to assess efficacy and safety of this triplet (irinotecan, 5FU/LV and oxaliplatin) in second-line treatment in fit patients (ECOG 0-1) metastatic PDAC.

The primary objective is to assess the efficacy of NALIRINOX (= investigational arm) and NALIRI (= standard care arm) in terms of Progression-Free Survival Rate (PFSR).

As secondary objectives, the following will be evaluated in both arms:

* Safety/toxicity and tolerability profile according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.
* Progression free survival (PFS)
* Overall response rate and duration of response as assessed by imaging (RECIST 1.1) and tumor markers
* Overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic adenocarcinoma of the pancreas
* Progression documented after gemcitabine-Abraxane, or gemcitabine monotherapy
* Signed written informed consent
* Age ≥ 18
* ECOG PS 0/1 at study entry
* Measurable disease
* Adequate renal (serum creatinine ≤ 1.5x upper reference range), liver (total bilirubin ≤ 1.5x upper reference range) and hematopoietic functions (PMN ≥ 1,5x109/L, platelets ≥ 100x109/L, hemoglobin ≥ 9g/dl)
* INR/PTT ≤ 1.5x ULN
* Life expectancy of at least 12 weeks
* Effective contraception for both male and female patients if the risk of conception exists during treatment and for one month after the last administration
* Peripheral Neuropathy < grade 2

Exclusion Criteria:

* Uncontrolled concurrent CNS, cardiac, infectious diseases, hypertension
* History of myocardial infarction, deep venous or arterial thrombosis, CVA during the last 6 months
* Known hypersensitivity to any of the components, including excipients, of study treatments
* Previous malignancy in the last past 3 years except basal cell cancer of the skin or preinvasive cancer of the cervix or carcinoma in situ of any type
* Pregnancy or breast feeding
* Medical or psychological conditions that would not permit the patient to complete the study or sign inform consent
* Unstable angina, congestive heart failure ≥NYHA class II
* Uncontrolled hypertension despite optimal management (systolic blood pressure >150 mmHg or diastolic pressure > 90mmHg)
* HIV infection
* Complete DPD deficiency
* Liver failure, cirrhosis Child Pugh B or C
* Active chronic hepatitis B or C with a need for antiviral treatment
* Brain metastasis
* Major surgery, open biopsy or significant traumatic injury within 4 weeks prior to the first dose of treatment
* History of organ allograft
* Ongoing uncontrolled, serious infection
* Renal failure requiring dialysis
* Patients receiving or having received any investigational treatment within 4 weeks prior to study entry, or participating to another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of NALIRINOX and NALIRI through Progression-Free Survival at D85 | at day 85 from randomization
  NALIRINOX is the investigational arm and NALIRI is the standard care arm. The efficacy will be assessed in terms of the Progression-Free Survival Rate (PFSR). This is defined as the proportion of patients alive and free of progression at day 85.

SECONDARY OUTCOMES:
Safety/toxicity and tolerability profil: Severety of adverse events | until 14 days after End of Treatment
  Adverse events and Serious Adverse events will be assessed during the study treatment and until 14 days later. Severety will be graded according to the NCI-CTCAE version 5.0 and relationship to the study medication will be defined.
Safety/toxicity and tolerability profil: Laboratory assessments | until 14 days after End of Treatment
  Standard laboratory safety assessments: They are mandatory prior to each administration of study medication and at the 15 days follow-up visit.
  Clinically significant vs not clinically significant.
Safety/toxicity and tolerability profil: ECOG | until 14 days after End of Treatment
  WHO ECOG performance status (PS) will be defined prior to each administration of study medication and at the 15 days follow-up visit following the ECOG Performance Status Scale.
Safety/toxicity and tolerability profil: review of body systems | until 14 days after End of Treatment
  A full review of body systems will be performed: heart rate, blood pressure, respiratory rate, body temperature, height, weight and ECG (screening visit only, unless clinically indicated).
  Clinically significant versus not clinically significant
Progression Free Survival and sensitivity analysis: Effect of Center on prognostic factors | From date of first study treatment administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years after End of Treatment.
  The effect of potential prognostic factors will be assessed through sensitivity analyses, including:
  * Investigational Center
Progression Free Survival and sensitivity analysis: Effect of tumor location on prognostic factors | From date of first study treatment administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years after End of Treatment
  The effect of potential prognostic factors will be assessed through sensitivity analyses, including:
  * Location of tumor (head of the pancreas versus other location)
Progression Free Survival and sensitivity analysis: Effect of previous chemotherapy on prognostic factors | From date of first study treatment administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years after End of Treatment
  The effect of potential prognostic factors will be assessed through sensitivity analyses, including:
  * Previous chemotherapy: gemcitabine alone vs gem-abx
Progression Free Survival and sensitivity analysis: effect of ECOG on prognostic factors | From date of first study treatment administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years after End of Treatment
  The effect of potential prognostic factors will be assessed through sensitivity analyses, including:
  * WHO ECOG performance status (0 versus 1)
Objective tumor response: Rate of complete response and partial response | performed within 28 days before start therapy, 3 times every 6 weeks and afterwards every 8 weeks
  Tumor (response) evaluation will be performed according to RECIST criteria v. 1.1 (CT scan thorax, abdomen and pelvis or MRI abdomen and pelvis + CT chest) based upon the investigator's assessment. Overall response is defined as a best response of either CR or PR (CR+PR).
Duration of overall survival | Time from Day 1 of therapy to death until maximum 5 years after End of Treatment
  For patients who are still alive at the time of study analysis or who are lost to follow up, survival will be censored at the last recorded date that the patient is known to be alive or at the date of data cut-off, whatever occurs earlier.
Duration of disease control | From date of first study treatment administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years after End of Treatment
  Disease control is defined as a best response of either CR, PR, or SD (CR+PR+SD).
Duration of response | Time from measurement criteria are first met for CR/PR to either the first time disease progression is documented or death (for not progressed patients who deceased within 60 days from last tumor assessment) until maximum 5 years after EOT
  The duration of response will be censored on the date of last known tumor assessment for not progressed patients lost to follow up or deceased prior to the next planned tumor assessment (within 60 days). Not evaluable patients at one time point assessment will be censored at the date of last known assessment.

OTHER OUTCOMES:
Exploratory lab investigation for potential prognostic and predictive biomarkers on blood and tumor samples | Sapmples will be collected throughout the study and shipped to the sponsor maximum 1 year after last 15 day follow-up visit
  Translational research will be performed for potential prognostic and predictive biomarkers. For that purpose, plasma samples will be kept in the selected centres' biobanks.
  The translational research will be carried out on tumor samples collected before the start of treatment and on blood samples collected as per below.
  Tumor tissue:
  10 slices of the paraffin embedded tissue collected during the diagnosis of the disease will be collected.
  Blood samples:
  Two 10 ml blood samples from each patient who consents to participate in the biological study will be collected before the start of the treatment, and before each cycle till the discontinuation of the treatment.
  The exact measurements that will be done, have not been defined yet.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borbath, Principal Investigator — University hospital St-luc, Brussel
Locations (13):
- Belgium (13):
  - UZ Antwerpen, Antwerp, Antwerp
  - ULB Erasme, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc UCL, Brussels, Brussels Capital
  - CHC MontLégia, Liège, Liège
  - AZ St-Lucas, Bruges, West-Vlaanderen
  - AZ Imelda, Bonheiden
  - Grand Hopital de Charleroi, Charleroi
  - AZ Maria Middelares, Ghent
  - University Hospital Ghent, Ghent
  - Pôle Hospitalier Jolimont (HELORA), Haine-Saint-Paul
  - CHU Ambroise Paré, Mons
  - CHR Namur, Namur
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No